CLINICAL TRIAL: NCT06678945
Title: Comparing Two Different Attachments Retaining Mandibular Implant Overdenture Regarding Retention and Patient Satisfaction (Randomized Clinical Trail)
Brief Title: Using Two Different Attachments in Mandibular Implant Overdenture Cases in Order to Retention and Patient Satisfaction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Noha Taha Kamel Taha Alloush, Lecturer, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27 4 24
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Edentulous Alveolar Ridge; Complete Edentulism; Dental Implant; Attachments; Implant Supported Overdenture; Edentulous Mouth; Edentulous Jaw
Keywords: Dental Implants; Completely edentulous patients; Edentulous Ridge
MeSH Terms: conditions — Mouth, Edentulous; Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bar-Clip attachment (Active Comparator): on the 2nd stage, implants will be loaded with bar-clip attachments to support overdenture
  Interventions: Procedure: Bar-Clip attachment
- Bar- OT Equator attachment (Experimental): on the 2nd stage, implants will be loaded with Bar- OT Equator attachments to support overdenture
  Interventions: Procedure: Bar- OT Equator attachment

INTERVENTIONS:
Procedure: Bar-Clip attachment — The 2 implants will be connected with bar attachments while the denture will be retained over the bar using clip.
  Arms: Bar-Clip attachment
Procedure: Bar- OT Equator attachment — The 2 implants will be connected with bar attachments while the denture will be retained over the bar using the OT Equator.
  Arms: Bar- OT Equator attachment

SUMMARY:
The Goal of the clinical trail is to evaluate the efficacy of Bar- OT Equator attachment on retention and patient satisfaction in comparison to the standard technique using Bar- clip attachment.

Patients will visit the clinic after the surgery and after the attachment insertion for check ups and during the follow up periods ( at denture insertion, 3 months and 6 months)

DETAILED DESCRIPTION:
patients will receive upper complete dentures and lower complete overdentures. The upper complete denture will be mucosa supported and the lower complete denture will be supported and retained for all patients by two dental implants in the inter-foraminal region. Patients will be divided into two equal groups; Group I will be retained by Bar-Clip attachment, while Group II will be retained by Bar- OT Equator attachment. Both groups will be functionally loaded after three months of insertion.

Retention of lower denture will be measured using digital force gauge and Patient satisfaction was evaluated with a standard 5-point Liker scale questionnaire. All parameters will be measured at denture insertion, 3 month, and 6 month later.

ELIGIBILITY:
Inclusion Criteria:

* All patients age must range from 60- 70 years old.
* All patients' ridges should be covered with firm mucosa free from any signs of inflammation or ulceration and exhibit adequate height and width of the residual alveolar ridge.
* Patients should be free from any metabolic or bone disorder that contraindicate implant installation.
* All patients must have sufficient inter arch space

Exclusion Criteria:

1. Patients with oral or systemic diseases.
2. Patients with xerostomia or excessive salivation.
3. Patients with parafunctional habits (bruxism or clenching).
4. Heavy smoker or alcoholic patients.
5. Patients with history of temporo-mandibular dysfunction.
6. Patients with brain disorders or psychiatric disorders

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Retention | it will be measured at denture insertion, 3 month, and 6 month later
  Retention will be measured using digital force gauge A digital force meter was used to measure denture resistance to vertical displacement (i.e., retention) by applying a pulling force on a metal hook located in the geometric center of each mandibular conventional denture that was identified on the lower cast at the intersection of three lines bisecting the angles of the triangle, formed by both retromolar pads and the midline.
  Measurement of mandibular denture retention:
  The patient was instructed to place his head on chin rest and occlusal plane was set parallel to the floor. Tongue freedom was checked then and three minutes seating time was allowed before taking the measurements. A vertical pulling force was applied using the metallic probe of the digital force-meter that was attached to the hook present at the geometric center of mandibular denture. Average value of six readings was recorded.

SECONDARY OUTCOMES:
Patient satisfaction | it will be measured at denture insertion, 3 month, and 6 month later.
  Patient satisfaction was evaluated with a standard 5-point Liker scale questionnaire, which included subjective parameters such as initial adaptability, post insertion problems, aesthetics, masticatory ability, speech, retention. Patients were asked to respond to questions given in the questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Al Saraya, Old Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Clinical Study Report
Supporting Information: Study Protocol, CSR
Time Frame: Start Date: After publication End Date: 10 years
Access Criteria: After publication through the corresponding author